CLINICAL TRIAL: NCT01975753
Title: First Evaluation of Morphine Hydrochloride by Nebulisation Compared to Intravenous Route in Healthy Volunteers: Preliminary Study Dose
Brief Title: First Evaluation of Morphine Hydrochloride by Nebulisation in Healthy Volunteers
Acronym: AEROMORPH1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/004/HP
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Acute Pain
Keywords: pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Morphine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous morphine (Active Comparator): one bolus of intravenous morphine
  Interventions: Drug: Morphine
- nebulized morphine (Experimental): one "nebulized" bolus of morphine
  Interventions: Drug: Morphine
- fentanyl (Active Comparator): one "nebulized" bolus of fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Morphine
  Arms: Intravenous morphine; nebulized morphine
Drug: Fentanyl
  Arms: fentanyl

SUMMARY:
Acute pain relief in emergency setting is still a public health priority. Pain is the primary reason for emergency room use, but the situation of "oligo-analgesia" persists in all countries. Intravenous morphine titration has become the standard method for severe acute pain management in the emergency department, but it is still insufficiently implemented. Deviations from the recommended protocol are common: initial additional loading doses, unusually extended intervals between bolus, premature discontinuation. Several factors contribute to these difficulties: heaviness of its setting up, especially in overcrowding case, procedure rigidity, high consumption of nursing time. This method requires a systematic intravenously route, which has several inconvenients: algogenic procedures, coupled initial diagnostic venous sampling (delay for analgesia), excessive "medicalization" of ambulatory patients (risk of infection and less mobility in the emergency department). An alternative to reduce the analgesic latency in emergency department, without losing the benefits of tolerance and safety should be welcome. The inhaled route looks promising, but has yet not been enough evaluated in adults, and even less in the emergency room. Aerosol techniques change from one study to another (molecules, materials, doses, painful intensities included, judgment criteria and assessment times). A morphine titration by aerosol therapy could be an interesting alternative to the standard method disadvantages, using faster, painless and easier procedures, leading to "demedicalization".

To the need for stronger fundamentals, an additional study was designed in healthy volunteers. The objective is to compare the titration of intravenous morphine titration aerosol in moderate acute pain caused by electrostimulation.

To purchase this aim, we first need to determine accurately the smallest dose of effective and well tolerated inhaled morphine, to provide the "bolus" dose we have to repeat by titration, which is still currently unknown. This dose is called ED50, it's the effective dose for at least 50% of healthy volunteers relieved. ED50 for intravenous morphine is also needed to be established, unknown in this indication. The determination of these two parallel ED50 would allow a reliable conversion factor between the two routes of administration for morphine "bolus", which can then be tested in comparative titrations. To validate our induced pain model in healthy volunteers, we also have chosen to fix in these conditions the ED50 of fentanyl that the effective dose by nebulization is better known. This study would also describe the pharmacokinetics of inhaled morphine and its derivatives after a single spray.

ELIGIBILITY:
Inclusion Criteria:

* Sex: We choose to include 50% of men and 50% women (this covariate will be included in the parameters to balance the randomization list).
* Age: Healthy volunteers will be between 18 to 60 years
* Body mass index (BMI) between 19 and 29 kg / m²
* effective contraception methods in women of childbearing age
* Signature of informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Taking painkillers long-term
* Taking psychotropic drugs long-term
* Healthy volunteers with chronic pain
* Drug addiction
* Chronic neuropsychiatric pathology which may alter the pain threshold
* Active Smoking
* Chronic obstructive or restrictive respiratory pathology
* Progressive known pathology (hypertension, kidney failure, heart, liver ...)
* Chronic treatments are prohibited except oral contraception
* Delirium or dementia, people who did not understand the pain scales
* Lack of understanding of the French language
* pregnancy and lactation
* Poor venous capital
* History of abnormal reaction at a local / regional anesthesia
* Heart rate : HR <50 bpm
* Hypotension TAsyst with systolic blood pressure <100 mm Hg
* Atrioventricular block (PR interval> 200 ms)
* Period exclusion of another biomedical research
* Nobody placed under judicial protection, guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Effective doses of intravenous morphine hydrochloride "bolus" and nebulized "bolus" in 50% of healthy painful volunteers | 7 min
  The primary endpoint is efficacy: relief from healthy volunteers thanks to VAS decreasing, defined as ≤ 20 (100mm). At the end of the study the dose chosen is the effective dose for 50% of the volunteers.

SECONDARY OUTCOMES:
safety | 7 min
  Check tolerance of aerosols on respiratory and systemically 2. Describe the pharmacokinetics of a "bolus" and a titration of morphine hydrochloride aerosol standardized, and of all its metabolites 3. Establish the concentration-effect relationship of a spray "bolus" and of a titration of morphine hydrochloride standardized (for the analgesic effect) using a pharmacokinetic / pharmacodynamic model (PK / PD) and mathematical modeling 4. Methodological validation by determining the ED50 of a inhaled fentanyl "bolus" 5. Establish pharmacokinetic bases that can provide a secure further study in the emergency room, targeting patients with severe spontaneous acute pain

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Rouen, Haute Normandie, France

REFERENCES:
- [Background] Lvovschi V, Aubrun F, Bonnet P, Bouchara A, Bendahou M, Humbert B, Hausfater P, Riou B. Intravenous morphine titration to treat severe pain in the ED. Am J Emerg Med. 2008 Jul;26(6):676-82. doi: 10.1016/j.ajem.2007.10.025. PMID 18606320
- [Derived] Blum CA, Velly L, Brochet C, Ziegler F, Tavolacci MP, Hausfater P, Lvovschi VE. Relevance of cortisol and copeptin blood concentration changes in an experimental pain model. Sci Rep. 2022 Mar 19;12(1):4767. doi: 10.1038/s41598-022-08657-4. PMID 35306524